CLINICAL TRIAL: NCT02535949
Title: Tranexamic Acid Mechanisms and Pharmacokinetics in Traumatic Injury (TAMPITI TRIAL)
Brief Title: Tranexamic Acid Mechanisms and Pharmacokinetics in Traumatic Injury
Acronym: TAMPITI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TAMPITI TRIAL
Record Dates: First submitted 2014-12-05; First posted 2015-08-31 (Estimated); Results first posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Hemorrhage; Shock; Wounds and Injuries
MeSH Terms: conditions — Hemorrhage; Shock; Wounds and Injuries | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tranexamic Acid 2 Gram (Experimental): One time dose IV TXA 2 Grams given over 10 minutes within 2 hours of initial injury
  Interventions: Drug: Tranexamic Acid
- Tranexamic Acid 4 Gram (Experimental): One time dose IV TXA 4 Grams given over 10 minutes within 2 hours of initial injury
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): Matching Volume Normal Saline Placebo given IV over 10 minutes within 2 hours of initial injury
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — Tranexamic acid is a man-made form of an amino acid (protein) called lysine. Tranexamic acid prevents enzymes in the body from breaking down blood clots.
  Other Names: Cyklokapron
  Arms: Tranexamic Acid 2 Gram; Tranexamic Acid 4 Gram
Other: Placebo — Matching Volume Normal Saline Placebo given IV over 10 minutes within 2 hours of initial injury
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of TXA on the immune system, its pharmacokinetics, as well as safety and efficacy in severely injured trauma patients.

DETAILED DESCRIPTION:
Trauma is the leading cause of death in persons younger than 40 years. Hemorrhage is the etiology in 30% of these deaths, and remains the leading cause of potentially preventable mortality (66-80%) on the battlefield. Death secondary to hemorrhagic shock occurs from both surgical bleeding and coagulopathy. Due to the knowledge of increased fibrinolysis promoting a hypocoagulable state in severe trauma, trials have been performed to determine if antifibrinolytics such as tranexamic acid (TXA) could reduce morbidity and mortality by reducing death from hemorrhage. TXA is an antifibrinolytic that inhibits both plasminogen activation and plasmin activity, thus preventing clot break-down rather than promoting new clot formation. Despite the extensive use of TXA in many surgical populations and an increasing use in severe trauma patients, TXA does not have an FDA approved indication for patients with traumatic injuries. The effect of TXA on immune function has not been thoroughly examined, especially in patients with severe traumatic injury. The study of the effects of TXA use on endothelial activation and injury is also important due to the inter-relationship between coagulation and endothelial function. Endothelial injury secondary to local hypoperfusion causes acute traumatic coagulopathy with fibrinolysis. Therefore a thorough and comprehensive evaluation of the effects of TXA on immune, coagulation, and endothelial parameters is important to allow for a better understanding of the mechanisms of action of this agent.

This is a randomized placebo controlled trial to obtain mechanism of action data, pharmacokinetic information, and efficacy and safety data for the use of TXA in severely injured trauma patients. Participants will be randomized into 1 of 3 treatment arms (1:1:1): TXA 2 gram IV bolus, TXA 4 gram IV bolus, or placebo. The study period is from time of enrollment to hospital discharge or transfer. The study intervention will occur only once upon enrollment in the trial. Participants will receive study drug within two hours from their initial injury. Blood samples will be drawn at multiple time points for immune parameters, Pharmacodynamics, and repository samples.

Immune parameter samples will be drawn at at approximately 0, 6, 24 and 72 hours after study drug/placebo administration.

Pharmacokinetic and pharmacodynamic samples will be drawn according to two schedules. Even number sampling times, blood will be drawn at the approximate time points: 0, 20 min, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, and 12 hr. A patient sampled on odd number sampling times will have samples drawn at the approximate time points: 0, 10 min, 40 min, 1.5 hr, 3 hr, 6 hr, 10 hr and 24 hr.

Repository samples will be drawn at approximate time points: 0, 1, 6, 24, and 72 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with traumatic injury that are ordered to receive at least 1 blood product and/or
2. Patients admitted to the Emergency Department with a traumatic injury and require immediate transfer to the operating room to control the bleeding
3. Able to receive the study drug within 2 hours from estimated time of injury **Please note that in circumstances where the patient initially met inclusion/exclusion criteria (i.e. received blood products in the ED before a full evaluation of their injuries is complete) but is later found to only have a soft tissue involved injury or does not have a traumatic bleeding source), the Investigator may determine that the patient should not be randomized into the trial and the patient should be considered a screen failure

Exclusion Criteria:

1. Patients known to be < 18 years of age
2. Suspected Acute MI or stroke(thromboembolic and/or hemorrhagic) on admission
3. Known inherited coagulation disorders
4. Known history of thromboembolic events (DVT, PE, MI, Stroke)

   • Please note that past medical history of hemorrhagic stroke is permitted, but not current admission with hemorrhagic stroke
5. Known history of seizures and/or seizure after injury/on admission related to this hospitalization
6. Suspected or known pregnancy
7. Known to be lactating
8. Suspected or known prisoners
9. Futile care
10. Known current state of immunosuppression (i.e. on high dose steroids, chemotherapeutics, etc.)
11. Unknown estimated time of injury 12). Patients wearing an "Opt Out" TAMPITI Study bracelet 13). Known presence of subarachnoid hemorrhage.

14.) Isolated injuries to hands and/or feet (distal) 15.) Administration of antifibrinolytics pre-hospital and/or during this ED admission prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-02; Primary Completion 2017-07-04 (Actual); Study Completion 2017-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip C Spinella, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Derived] Spinella PC, Thomas KA, Turnbull IR, Fuchs A, Bochicchio K, Schuerer D, Reese S, Coleoglou Centeno AA, Horn CB, Baty J, Shea SM, Meledeo MA, Pusateri AE, Levy JH, Cap AP, Bochicchio GV; TAMPITI Investigators. The Immunologic Effect of Early Intravenous Two and Four Gram Bolus Dosing of Tranexamic Acid Compared to Placebo in Patients With Severe Traumatic Bleeding (TAMPITI): A Randomized, Double-Blind, Placebo-Controlled, Single-Center Trial. Front Immunol. 2020 Sep 8;11:2085. doi: 10.3389/fimmu.2020.02085. eCollection 2020. PMID 33013880

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tranexamic Acid 2 Gram | Tranexamic Acid 4 Gram | Placebo
Started | 50 | 50 | 50
Completed | 49 | 50 | 50
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All analysis is based on the number of participants per group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid 2 Gram | Tranexamic Acid 4 Gram | Placebo | Total
Number analyzed (Participants) | 49 | 50 | 50 | 149
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 0 | 2
  Between 18 and 65 years | 47 | 46 | 49 | 142
  >=65 years | 1 | 3 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 5 | 18
  Male | 44 | 42 | 45 | 131
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 42 | 43 | 44 | 129
  White | 7 | 6 | 5 | 18
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 49 | 50 | 50 | 149

OUTCOME MEASURES:

1. Primary Outcome: Change in HLA-DR Expression on Monocytes 72 Hours After Drug or Placebo Administration in Patient Groups (0g TXA (Placebo); 2g TXA; 4g TXA)."
Description: Blood was drawn from patients at baseline (0 h, just before placebo or drug administration) and at 72 hours post placebo or drug administration. Leukocytes in these blood samples were stained with fluroescent antibodies specific for CD45, CD14, and HLA-DR, analyzed by flow cytometry, and the median fluorescen intensity (MFI) of HLA-DR signal was recorded for monocytes (CD45+CD14+). The fold change in HLA-DR expression from prior to placebo/drug administration to 72 h after placebo/drug administration ("0 h : 72 h") was calculated as HLA-DR MFI72hours ÷ HLA-DR CD14 MFI0hours. Non-paramteric one-way ANOVA (Kruskal-Wallis test) was performed between each treatment group at the given time pont, and the p-value reported.
Time Frame: Samples Drawn through 72 hours after study initiation
Population: Change in HLA-DR Expression on Monocytes 72 hours after administration. Leukocytes stained with antibodies and analyzed by flow cytometry. The median fluorescen intensity of HLA-DR signal was measured for monocytes at 0 and 72 hours. Non-paramteric one-way ANOVA was performed and the p-value reported.
Measure: Median (Inter-Quartile Range); unit: fold change
Arm/Group | Tranexamic Acid 2 Gram | Tranexamic Acid 4 Gram | Placebo
Number analyzed (Participants) | 49 | 50 | 50
fold change | 0.503 [0 to 0.717] | 0.509 [0.336 to 0.733] | 0.532 [0.371 to 0.736]

2. Secondary Outcome: Differences in Cytokine Profiles Between the Three Study Groups
Description: To evaluate the effects of TXA on immune function parameters we will, in a RCT, analyze samples from 150 patients (50 in each study group), at multiple time points. Parameters are:
  a. Cytokines measured from time 0 to 72 hours.
Time Frame: Samples Drawn through 72 hours after study initiation
Population: Cytokine Levels at 0 and 72 hours after drug or placebo administration in patient groups. Blood was drawn, serum isolated, and frozen. Frozen sera were thawed and the listed cytokines measured uisng a multiplexed platform. Non-paramteric one-way ANOVA was performed between each treatment group, and the p- value reported.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Tranexamic Acid 2 Gram | Tranexamic Acid 4 Gram | Placebo
Number analyzed (Participants) | 49 | 50 | 50
pg/mL
  ITAC hour 0 | 34.24 [25.02 to 55.19] | 32.75 [21.34 to 49.41] | 29.34 [17.92 to 44.44]
  ITAC hour 72 | 25.67 [20.76 to 41.14] | 21.69 [13.98 to 34.58] | 21.58 [13.8 to 33.24]
  GM-CSF hour 0 | 67.79 [46.73 to 111.19] | 67.58 [43.91 to 125.74] | 64.69 [39.83 to 97.43]
  GM-CSF hour 72 | 69.22 [34.07 to 107.56] | 52.88 [38.41 to 94.83] | 61.41 [46.09 to 96.77]
  Factalkine hour 0 | 223.61 [94.4 to 328.9] | 146.23 [103.15 to 210.32] | 141.8 [75.83 to 223.7]
  Factalkine hour 72 | 174.91 [116.22 to 239.2] | 124.23 [83.71 to 183.81] | 100.51 [74.7 to 187.04]
  IFNgamma hour 0 | 23.46 [13.25 to 38.08] | 17.59 [14.16 to 38.95] | 17.47 [9.49 to 25.81]
  IFNgamma hour 72 | 17.89 [12.22 to 30.44] | 14.79 [10.89 to 29.69] | 12.98 [9.06 to 28.48]
  IL-10 hour 0 | 115.98 [41.93 to 235.6] | 84.39 [46.77 to 127.73] | 105.07 [39.75 to 250.02]
  IL-10 hour 72 | 31.76 [14.47 to 46.13] | 42.39 [16.48 to 64.75] | 32.38 [19.7 to 44.71]
  MIP-3a hour 0 | 22.95 [14.03 to 29.38] | 21.94 [17.4 to 27.98] | 22.95 [12.36 to 31.03]
  MIP-3a hour 72 | 38.49 [23.43 to 132.02] | 27.61 [23.66 to 54.31] | 31.54 [17.89 to 50.33]
  IL-12p70 hour 0 | 9.5 [6.81 to 17.61] | 8.64 [6.04 to 12.65] | 8.78 [4.89 to 13.58]
  IL-12p70 hour 72 | 9.67 [5.86 to 14.06] | 9.45 [5.72 to 11.9] | 7.58 [3.78 to 17.51]
  IL-13 hour 0 | 11.8 [5.7 to 26.86] | 11.11 [5.37 to 23.82] | 9.08 [5.31 to 16.27]
  IL-13 hour 72 | 11.11 [5.78 to 27.37] | 10.27 [5.24 to 20.28] | 10.28 [4.42 to 18.9]
  IL -17A hour 0 | 21.51 [11.46 to 30.35] | 15.05 [9.9 to 24.01] | 18.73 [11.45 to 28.43]
  IL-17A hour 72 | 20.06 [11 to 38.72] | 16.67 [11.07 to 26.89] | 14 [9.35 to 29.42]
  IL-1beta hour 0 | 4.17 [2.49 to 6.63] | 3.75 [2.75 to 6.11] | 3.9 [2.77 to 5.7]
  IL-1beta hour 72 | 4.15 [2.75 to 5.34] | 3.44 [2.32 to 4.77] | 3.11 [2.4 to 6.01]
  IL-2 hour 0 | 4.17 [2.82 to 7.36] | 4.29 [2.62 to 7.07] | 4.01 [3.05 to 5.63]
  IL-2 hour 72 | 4.26 [2.4 to 8.62] | 3.49 [2.21 to 5.77] | 4.12 [2.74 to 7.07]
  IL-21 hour 0 | 6.28 [3.51 to 9.74] | 6.13 [3.64 to 9.75] | 7.02 [3.22 to 10.96]
  IL-21 hour 72 | 6.44 [3.89 to 13.59] | 6.95 [3.61 to 9.5] | 5.51 [2.79 to 10.92]
  IL-4 hour 0 | 69.45 [45.42 to 94.71] | 58.24 [41.97 to 79.64] | 58.16 [37.97 to 95.79]
  IL-4 hour 72 | 49.99 [29.39 to 73.91] | 40.5 [24.45 to 75.08] | 35.53 [23.24 to 68.29]
  IL-23 hour 0 | 724.45 [445.25 to 1105.5] | 428.26 [244.36 to 875.62] | 406.46 [244.04 to 773.56]
  IL-23 hour 72 | 589.73 [388.72 to 893.66] | 351.47 [258.99 to 811.79] | 399.74 [248.94 to 971.77]
  IL-5 hour 0 | 9.3 [4.12 to 15.79] | 9.48 [5.17 to 15.28] | 9.06 [5.72 to 13.27]
  IL-5 hour 72 | 8.68 [6.31 to 17.87] | 8.05 [6.12 to 15.22] | 8.32 [6.94 to 13.44]
  IL-6 hour 0 | 54.48 [23 to 182.07] | 39.7 [18.27 to 97.99] | 63.56 [28.05 to 110.6]
  IL-6 hour 72 | 73.97 [35.27 to 156.11] | 67.95 [32.83 to 149.24] | 41.9 [21.71 to 70.01]
  IL-7 hour 0 | 18.53 [12.67 to 30.56] | 15.33 [11.47 to 24.3] | 16.52 [10.19 to 23.65]
  IL-7 hour 72 | 18.47 [11.19 to 27.49] | 16.24 [11 to 22.19] | 16.8 [10.93 to 19.66]
  IL-8 hour 0 | 15.25 [10.43 to 31.68] | 13.59 [9.62 to 24.65] | 13.78 [8.03 to 26.45]
  IL-8 hour 72 | 26.9 [18 to 42.11] | 23.05 [17.14 to 38.97] | 17.64 [13.78 to 23.71]
  MIP-1alpha hour 0 | 32.57 [22.77 to 42.48] | 30.98 [20.36 to 42.9] | 27.85 [21.99 to 41.89]
  MIP-1alpha hour 72 | 28.57 [20.69 to 43.98] | 27.24 [18.05 to 39.23] | 25.47 [17.29 to 43.96]
  MIP-beta hour 0 | 44.91 [31.8 to 54.57] | 37.66 [13.55 to 48.35] | 35.44 [24.74 to 50.11]
  MIP-beta hour 72 | 36.78 [25.72 to 45.65] | 29.02 [23.15 to 39.4] | 28.15 [22.23 to 36.19]
  TNFa hour 0 | 19.16 [13.34 to 23.46] | 16.4 [13.3 to 20.5] | 16.4 [12.3 to 21.17]
  TNFa hour 72 | 19.38 [17.57 to 25.85] | 20.09 [15.82 to 25.62] | 16.16 [12.37 to 21.36]

3. Secondary Outcome: Differences in Leukocyte Function Parameters Between the Three Study Groups
Description: To evaluate the effects of TXA on immune function parameters we will, in a RCT, analyze samples from 150 patients (50 in each study group), at multiple time points. Parameters are:
  a. Flow cytometric analyses on leukocytes measured from time 0 to 72 hours.
Time Frame: Samples Drawn through 72 hours after study initiation
Population: Change in CD11b and CD16 Expression on neutrophils 72 hours after. Leukocytes stained with antibodies specific and analyzed by flow cytometry. The median fluorescen intensity of CD11b or CD16 signal was measured on neutrophils. The fold change was measured, MFI72hours/MFI0hours. Non-paramteric one-way ANOVA was performed and the p-value reported.
Measure: Median (Inter-Quartile Range); unit: Fold Change
Arm/Group | Tranexamic Acid 2 Gram | Tranexamic Acid 4 Gram | Placebo
Number analyzed (Participants) | 49 | 50 | 50
Fold Change
  CD 11b+ | 0.875 [0.667 to 1.11] | 0.967 [0.802 to 1.207] | 0.844 [0.713 to 1.02]
  CD 16+ | 0.917 [0.733 to 0.994] | 0.870 [0.731 to 0.994] | 0.817 [0.703 to 0.942]

4. Secondary Outcome: Total Transfusion Volume CL
Description: Pharmacokinetic data was analyzed with NONMEM, using both the first-order and conditional non-Laplacian (with centering) estimation techniques. We considered two- and three-compartment models, parameterized in terms of both compartment volumes and clearances (distribution and elimination). We compared a basic model (in which pharmacokinetic parameters were independent of weight) to a model in which the pharmacokinetic parameters were assumed to be proportional to weight. The optimal model was selected on the basis of the objective function logarithm of the likelihood of the results) using standard criteria (NONMEM guide).
  Equations from optimal model:
  CL=109*((WT/70)**0.75) * (SCRint^-0.084) * ((NIRSInt)/96)^ -0.27 ) * ((PLTint)/130)^0.45) V1=1,160*(WT/70) * (TxTot)^0.03) Q=174*((WT/70)**0.75) V2=1080 *(WT/70)
  "Total Transfusion Volume CL" equals clearance (CL) affected by the covariate of Total Transfusion Volume (TxTot). This value is unitless per NONMEM reporting.
Time Frame: 24 hours
Population: Of the 99 participants analyzed, 49 received the 2 gram dose and 50 received the 4 gram dose.
Measure: Mean (95% Confidence Interval); unit: unitless
Groups:
- Tranexamic Acid 2 Gram and 4 Gram: One time dose IV TXA 2 Grams or 4 Grams given over 10 minutes within 2 hours of initial injury
  Tranexamic Acid: Tranexamic acid is a man-made form of an amino acid (protein) called lysine. Tranexamic acid prevents enzymes in the body from breaking down blood clots.
Arm/Group | Tranexamic Acid 2 Gram and 4 Gram
Number analyzed (Participants) | 99
unitless | 0.03 [0.007 to 0.05]

5. Secondary Outcome: Determine the Incidence of Thromboembolic Events (DVT, MI, PE, Stroke) in All Three Study Groups.
Description: The number of events per group for the incidence of thromboembolic events (DVT, MI, PE, Stroke) in all three study groups.
Time Frame: Hospital Discharge (average 10 days)
Population: The incidence of thromboembolic events (DVT, MI, PE, Stroke) in all three study groups are given based on events per group.
Measure: Number; unit: events
Arm/Group | Tranexamic Acid 2 Gram | Tranexamic Acid 4 Gram | Placebo
Number analyzed (Participants) | 49 | 50 | 50
events | 13 | 16 | 6

6. Secondary Outcome: Determine the Incidence of Seizures at 24 Hours in All Three Study Groups.
Description: The incidence of seizures at 24 hours in all three study groups. Number of participants with seizures are reported
Time Frame: 24 hours following TXA
Population: The incidence of seizures at 24 hours in all three study groups. This was done by totaling the number of participants with reported seizures.
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid 2 Gram | Tranexamic Acid 4 Gram | Placebo
Number analyzed (Participants) | 49 | 50 | 50
Participants | 0 | 1 | 0

7. Secondary Outcome: Determine the Incidence of All Adverse Events in All Three Study Groups
Description: All adverse events were totaled for each of the three study groups based on the number of incidents.
Time Frame: Hospital Discharge (average 10 days)
Population: The number of incidents were totaled for the three study groups.
Measure: Number; unit: events
Arm/Group | Tranexamic Acid 2 Gram | Tranexamic Acid 4 Gram | Placebo
Number analyzed (Participants) | 49 | 50 | 50
events | 168 | 264 | 138

8. Secondary Outcome: Platelet Count CL
Description: Pharmacokinetic data was analyzed with NONMEM, using both the first-order and conditional non-Laplacian (with centering) estimation techniques. We considered two- and three-compartment models, parameterized in terms of both compartment volumes and clearances (distribution and elimination). We compared a basic model (in which pharmacokinetic parameters were independent of weight) to a model in which the pharmacokinetic parameters were assumed to be proportional to weight. The optimal model was selected on the basis of the objective function logarithm of the likelihood of the results) using standard criteria (NONMEM guide).
  Equations from optimal model:
  CL=109*((WT/70)**0.75) * (SCRint^-0.084) * ((NIRSInt)/96)^ -0.27 ) * ((PLTint)/130)^0.45) V1=1,160*(WT/70) * (TxTot)^0.03) Q=174*((WT/70)**0.75) V2=1080 *(WT/70)
  "Platelet Count CL" equals clearance (CL) affected by the covariate of Platelet Count (PLTint). This value is unitless per NONMEM reporting.
Time Frame: 24 hours
Population: Of the 99 participants analyzed, 49 received the 2 gram dose and 50 received the 4 gram dose.
Measure: Mean (95% Confidence Interval); unit: unitless
Arm/Group | Tranexamic Acid 2 Gram and 4 Gram
Number analyzed (Participants) | 99
unitless | 0.45 [0.28 to 0.61]

9. Secondary Outcome: Near Infrared Spectroscopy CL
Description: Pharmacokinetic data was analyzed with NONMEM, using both the first-order and conditional non-Laplacian (with centering) estimation techniques. We considered two- and three-compartment models, parameterized in terms of both compartment volumes and clearances (distribution and elimination). We compared a basic model (in which pharmacokinetic parameters were independent of weight) to a model in which the pharmacokinetic parameters were assumed to be proportional to weight. The optimal model was selected on the basis of the objective function logarithm of the likelihood of the results) using standard criteria (NONMEM guide).
  Equations from optimal model:
  CL=109*((WT/70)**0.75) * (SCRint^-0.084) * ((NIRSInt)/96)^ -0.27 ) * ((PLTint)/130)^0.45) V1=1,160*(WT/70) * (TxTot)^0.03) Q=174*((WT/70)**0.75) V2=1080 *(WT/70)
  "Near Infrared Spectroscopy CL" equals clearance (CL) affected by the covariate of Near Infrared Spectroscopy (NIRSint). This value is unitless per NONMEM reporting.
Time Frame: 24 hours
Population: Of the 99 participants analyzed, 49 received the 2 gram dose and 50 received the 4 gram dose.
Measure: Mean (95% Confidence Interval); unit: unitless
Arm/Group | Tranexamic Acid 2 Gram and 4 Gram
Number analyzed (Participants) | 99
unitless | -0.27 [-0.38 to -0.15]

10. Secondary Outcome: Creatinine Count CL
Description: Pharmacokinetic data was analyzed with NONMEM, using both the first-order and conditional non-Laplacian (with centering) estimation techniques. We considered two- and three-compartment models, parameterized in terms of both compartment volumes and clearances (distribution and elimination). We compared a basic model (in which pharmacokinetic parameters were independent of weight) to a model in which the pharmacokinetic parameters were assumed to be proportional to weight. The optimal model was selected on the basis of the objective function logarithm of the likelihood of the results) using standard criteria (NONMEM guide).
  Equations from optimal model:
  CL=109*((WT/70)**0.75) * (SCRint^-0.084) * ((NIRSInt)/96)^ -0.27 ) * ((PLTint)/130)^0.45) V1=1,160*(WT/70) * (TxTot)^0.03) Q=174*((WT/70)**0.75) V2=1080 *(WT/70)
  "Creatinine Count CL" equals clearance (CL) affected by the covariate of Creatinine levels (SCRint). This value is unitless per NONMEM reporting.
Time Frame: 24 hours
Population: Of the 99 participants analyzed, 49 received the 2 gram dose and 50 received the 4 gram dose.
Measure: Mean (95% Confidence Interval); unit: unitless
Arm/Group | Tranexamic Acid 2 Gram and 4 Gram
Number analyzed (Participants) | 99
unitless | -0.084 [-0.13 to -0.03]

11. Secondary Outcome: V2- Peripheral Volume (L/70kg)
Description: Pharmacokinetic data was analyzed with NONMEM, using both the first-order and conditional non-Laplacian (with centering) estimation techniques. We considered two- and three-compartment models, parameterized in terms of both compartment volumes and clearances (distribution and elimination). We compared a basic model (in which pharmacokinetic parameters were independent of weight) to a model in which the pharmacokinetic parameters were assumed to be proportional to weight. The optimal model was selected on the basis of the objective function logarithm of the likelihood of the results) using standard criteria (NONMEM guide).
  Equations from optimal model:
  CL=109*((WT/70)**0.75) * (SCRint^-0.084) * ((NIRSInt)/96)^ -0.27 ) * ((PLTint)/130)^0.45) V1=1,160*(WT/70) * (TxTot)^0.03) Q=174*((WT/70)**0.75) V2=1080 *(WT/70)
  "V2" equals Peripheral Volume in L/70kg.
Time Frame: 24 hours
Population: Of the 99 participants analyzed 49 received the 2 gram dose and 50 received the 4 gram dose.
Measure: Mean (95% Confidence Interval); unit: L/70kg
Arm/Group | Tranexamic Acid 2 Gram and 4 Gram
Number analyzed (Participants) | 99
L/70kg | 1080 [959 to 1200]

12. Secondary Outcome: Q- Intercompartmental Clearance (L/70kg)
Description: Pharmacokinetic data was analyzed with NONMEM, using both the first-order and conditional non-Laplacian (with centering) estimation techniques. We considered two- and three-compartment models, parameterized in terms of both compartment volumes and clearances (distribution and elimination). We compared a basic model (in which pharmacokinetic parameters were independent of weight) to a model in which the pharmacokinetic parameters were assumed to be proportional to weight. The optimal model was selected on the basis of the objective function logarithm of the likelihood of the results) using standard criteria (NONMEM guide).
  Equations from optimal model:
  CL=109*((WT/70)**0.75) * (SCRint^-0.084) * ((NIRSInt)/96)^ -0.27 ) * ((PLTint)/130)^0.45) V1=1,160*(WT/70) * (TxTot)^0.03) Q=174*((WT/70)**0.75) V2=1080 *(WT/70)
  "Q" equals intercompartmental clearance in L/70kg.
Time Frame: 24 hours
Population: Of the 99 participants analyzed, 49 received the 2 gram dose and 50 received the 4 gram dose.
Measure: Mean (95% Confidence Interval); unit: L/70kg
Arm/Group | Tranexamic Acid 2 Gram and 4 Gram
Number analyzed (Participants) | 99
L/70kg | 174 [128 to 220]

13. Secondary Outcome: V1- Central Volume (L/70kg)
Description: Pharmacokinetic data was analyzed with NONMEM, using both the first-order and conditional non-Laplacian (with centering) estimation techniques. We considered two- and three-compartment models, parameterized in terms of both compartment volumes and clearances (distribution and elimination). We compared a basic model (in which pharmacokinetic parameters were independent of weight) to a model in which the pharmacokinetic parameters were assumed to be proportional to weight. The optimal model was selected on the basis of the objective function logarithm of the likelihood of the results) using standard criteria (NONMEM guide).
  Equations from optimal model:
  CL=109*((WT/70)**0.75) * (SCRint^-0.084) * ((NIRSInt)/96)^ -0.27 ) * ((PLTint)/130)^0.45) V1=1,160*(WT/70) * (TxTot)^0.03) Q=174*((WT/70)**0.75) V2=1080 *(WT/70)
  "V1" equals central volume in L/70kg.
Time Frame: 24 hours
Population: Of the 99 participants analyzed, 49 received the 2 gram dose and 50 received the 4 gram dose.
Measure: Mean (95% Confidence Interval); unit: L/70kg
Arm/Group | Tranexamic Acid 2 Gram and 4 Gram
Number analyzed (Participants) | 99
L/70kg | 1160 [968 to 1350]

14. Secondary Outcome: CL- Clearance of TXA (mL/(Min*70kg))
Description: Pharmacokinetic data was analyzed with NONMEM, using both the first-order and conditional non-Laplacian (with centering) estimation techniques. We considered two- and three-compartment models, parameterized in terms of both compartment volumes and clearances (distribution and elimination). We compared a basic model (in which pharmacokinetic parameters were independent of weight) to a model in which the pharmacokinetic parameters were assumed to be proportional to weight. The optimal model was selected on the basis of the objective function logarithm of the likelihood of the results) using standard criteria (NONMEM guide).
  Equations from optimal model:
  CL=109*((WT/70)**0.75) * (SCRint^-0.084) * ((NIRSInt)/96)^ -0.27 ) * ((PLTint)/130)^0.45) V1=1,160*(WT/70) * (TxTot)^0.03) Q=174*((WT/70)**0.75) V2=1080 *(WT/70)
  "CL" equals clearance of TXA in mL/(min*70kg).
Time Frame: 24 hours
Population: Of the 99 participants analyzed, 49 received the 2 gram dose and 50 received the 4 gram dose.
Measure: Mean (95% Confidence Interval); unit: mL/(min*70kg)
Arm/Group | Tranexamic Acid 2 Gram and 4 Gram
Number analyzed (Participants) | 99
mL/(min*70kg) | 109 [100 to 118]

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Tranexamic Acid 2 Gram | Tranexamic Acid 4 Gram | Placebo
All-Cause Mortality (participants affected / at risk) | 5/49 | 4/50 | 9/50
Serious Adverse Events (participants affected / at risk) | 14/49 | 18/50 | 13/50
Other Adverse Events (participants affected / at risk) | 25/49 | 39/50 | 26/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tranexamic Acid 2 Gram (N=49) | Tranexamic Acid 4 Gram (N=50) | Placebo (N=50)
Deep Vein Thrombosis (Vascular disorders) | 5 | 7 | 1
acute blood loss/anemia (Blood and lymphatic system disorders) | 2 | 2 | 1
Acute desaturation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 3 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Anastomatic Bleeding (Blood and lymphatic system disorders) | 0 | 2 | 0
Arterial Bleeding (Blood and lymphatic system disorders) | 2 | 0 | 0
Death (Injury, poisoning and procedural complications) | 4 | 3 | 9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tranexamic Acid 2 Gram (N=49) | Tranexamic Acid 4 Gram (N=50) | Placebo (N=50)
Pain (Injury, poisoning and procedural complications) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 6 | 16 | 6
Sepsis (Infections and infestations) | 6 | 6 | 2
Hypotension (Cardiac disorders) | 4 | 3 | 6
Anemia (Blood and lymphatic system disorders) | 8 | 9 | 8
Urinary tract infection (Infections and infestations) | 1 | 1 | 2
SVT (Cardiac disorders) | 0 | 2 | 0
Hyperphosphatemia (Blood and lymphatic system disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-17): https://cdn.clinicaltrials.gov/large-docs/49/NCT02535949/Prot_SAP_000.pdf